CLINICAL TRIAL: NCT02320838
Title: Unmodulated 5 Kilohertz Alternating Currents Versus TENS: Effect on Mechanical and Thermal Pain Thresholds, Tactile Threshold, and Peripheral Nerve Conduction in Humans.
Brief Title: Unmodulated 5 Kilohertz Currents Versus TENS: Effect on Pain Thresholds, Tactile Threshold, and Nerve Conduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Hospital Nacional de Parapléjicos de Toledo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: javendano
Record Dates: First submitted 2014-11-18; First posted 2014-12-19 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Pain
Keywords: Transcutaneous Electric Nerve Stimulation; Electric Stimulation Therapy; Unmodulated Alternating Currents; Neural Conduction; Pain Threshold
MeSH Terms: conditions — Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 5 KHz (Experimental): Transcutaneous application of 5 KHz current over the course of the superficial radial nerve in the right forearm for a 20 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold.
  Interventions: Device: 5 KHz
- TENS (Experimental): Transcutaneous application of Conventional TENS current over the course of the superficial radial nerve in the right forearm for a 20 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold. Currents parameters are frequency 110 Hz and pulse width 200 microseconds
  Interventions: Device: TENS
- Sham Stimulation (Sham Comparator): Electrodes are placed over the course of the superficial radial nerve in the right forearm for a 20 minutes in the same manner as experimental groups, but will be applied a sham electrical stimulation increasing the current intensity of an unconnected channel.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: 5 KHz — 5 KHz transcutaneous electrical stimulation over superficial radial nerve through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Arms: 5 KHz
Device: TENS — TENS transcutaneous electrical stimulation over superficial radial nerve through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Arms: TENS
Device: Sham stimulation — Sham transcutaneous electrical stimulation over superficial radial nerve through the electrotherapy device Myomed 932. (Enraf-Nonius, Delft, Netherlands)
  Arms: Sham Stimulation

SUMMARY:
The purpose of this study is to determine whether the transcutaneous application of unmodulated 5 Kilohertz (KHz) alternating currents are effective in decreasing the thermal and mechanical experimental pain and cause changes in peripheral nerve conduction. Moreover evidence whether the effect and comfort of this current is greater than Conventional TENS (Transcutaneous Electrical Nerve Stimulation) commonly used for the treatment of clinical pain.

DETAILED DESCRIPTION:
In the last years several animal experimental studies have evidenced that high frequency unmodulated currents about 5 KHz can cause a peripheral nerve block. However electric currents with these high frequencies that are usually used for the treatment of pain in humans are interrupted or modulated (i.e. interferential currents)

This evidences in animals could have application in pain treatment, characterized by overactive nervous system. For this reason it was decided to compare the effects on experimental pain and peripheral nerve conduction of this new electric current versus sham stimulation and TENS (Transcutaneous Electrical Nerve Stimulation).

The scientific literature on transcutaneous electrical stimulation in humans and changes in nerve conduction and / or somatosensory thresholds focuses mainly on TENS (Transcutaneous Electrical Nerve Stimulation). Therefore TENS is a good reference standard to compare the effect of this new currents.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be volunteer healthy students of Physiotherapy, University of Castilla - La Mancha, older than 18 years.

Exclusion Criteria:

* Neuromuscular disease.
* Epilepsy.
* Trauma, surgery or pain affecting the upper limb, shoulder girdle or cervical area.
* Osteosynthesis material in the upper limb.
* Diabetes.
* Cancer.
* Cardiovascular disease.
* Pacemaker or other implanted electrical device.
* Take any drug (NSAIDs, corticosteroids, antidepressants, analgesics, antiepileptics, ...) during the study and in the previous 7 days.
* Presence of tattoos or other external agent introduced into the treatment or assessment area.
* Pregnancy.
* Sensitivity disturbance in upper limb.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2014-11; Primary Completion 2015-01 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Avendaño-Coy, MsC, Principal Investigator — University of Castilla-La Mancha, Toledo, Spain

REFERENCES:
- [Derived] Avendano-Coy J, Gomez-Soriano J, Goicoechea-Garcia C, Basco-Lopez JA, Taylor J. Effect of Unmodulated 5-kHz Alternating Currents Versus Transcutaneous Electrical Nerve Stimulation on Mechanical and Thermal Pain, Tactile Threshold, and Peripheral Nerve Conduction: A Double-Blind, Placebo-Controlled Crossover Trial. Arch Phys Med Rehabil. 2017 May;98(5):888-895. doi: 10.1016/j.apmr.2016.11.020. Epub 2016 Dec 23. PMID 28017706

RESULTS

PARTICIPANT FLOW:
Groups:
- 5 KHz First, Then TENS and Then Sham; 5 KHz First, Then Sham and Then TENS: 5KHz: Transcutaneous application of 5 KHz current over the course of the superficial radial nerve in the right forearm for a 20 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold.
  TENS: Transcutaneous application of Conventional TENS current over the course of the superficial radial nerve in the right forearm for a 20 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold. Currents parameters are frequency 110 Hz and pulse width 200 microseconds.
  Sham Stimulation: Electrodes are placed over the course of the superficial radial nerve in the right forearm for a 20 minutes in the same manner as experimental groups, but will be applied a sham electrical stimulation increasing the current intensity of an unconnected channel.
- TENS First, Then 5 KHz and Then Sham: TENS: Transcutaneous application of Conventional TENS current over the course of the superficial radial nerve in the right forearm for a 20 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold. Currents parameters are frequency 110 Hz and pulse width 200 microseconds
  5KHz: Transcutaneous application of 5 KHz current over the course of the superficial radial nerve in the right forearm for a 20 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold.
  Sham Stimulation: Electrodes are placed over the course of the superficial radial nerve in the right forearm for a 20 minutes in the same manner as experimental groups, but will be applied a sham electrical stimulation increasing the current intensity of an unconnected channel.
- Sham First, Then TENS and Then 5KHz: Sham stimulation: Electrodes are placed over the course of the superficial radial nerve in the right forearm for a 20 minutes in the same manner as experimental groups, but will be applied a sham electrical stimulation increasing the current intensity of an unconnected channel.
  TENS: Transcutaneous application of Conventional TENS current over the course of the superficial radial nerve in the right forearm for a 20 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold. Currents parameters are frequency 110 Hz and pulse width 200 microseconds
  5KHz: Transcutaneous application of 5 KHz current over the course of the superficial radial nerve in the right forearm for a 20 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold.
- TENS First, Then Sham and Then 5KHz: ENS: Transcutaneous application of Conventional TENS current over the course of the superficial radial nerve in the right forearm for a 20 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold. Currents parameters are frequency 110 Hz and pulse width 200 microseconds
  5KHz: Transcutaneous application of 5 KHz current over the course of the superficial radial nerve in the right forearm for a 20 minutes session. The intensity of the current will increase until participants report a "strong but comfortable" sensation, just below motor threshold.
  Sham Stimulation: Electrodes are placed over the course of the superficial radial nerve in the right forearm for a 20 minutes in the same manner as experimental groups, but will be applied a sham electrical stimulation increasing the current intensity of an unconnected channel.
Period: First Intervention (1 Day)
Arm/Group | 5 KHz First, Then TENS and Then Sham | TENS First, Then 5 KHz and Then Sham | Sham First, Then TENS and Then 5KHz | TENS First, Then Sham and Then 5KHz | 5 KHz First, Then Sham and Then TENS
Started | 8 | 8 | 8 | 7 | 7
Completed | 8 | 8 | 8 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Washout (1 Day)
Arm/Group | 5 KHz First, Then TENS and Then Sham | TENS First, Then 5 KHz and Then Sham | Sham First, Then TENS and Then 5KHz | TENS First, Then Sham and Then 5KHz | 5 KHz First, Then Sham and Then TENS
Started | 8 | 8 | 8 | 7 | 7
Completed | 8 | 8 | 8 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | 5 KHz First, Then TENS and Then Sham | TENS First, Then 5 KHz and Then Sham | Sham First, Then TENS and Then 5KHz | TENS First, Then Sham and Then 5KHz | 5 KHz First, Then Sham and Then TENS
Started | 8 | 8 | 8 | 7 | 7
Completed | 8 | 8 | 8 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Washout (1 Day)
Arm/Group | 5 KHz First, Then TENS and Then Sham | TENS First, Then 5 KHz and Then Sham | Sham First, Then TENS and Then 5KHz | TENS First, Then Sham and Then 5KHz | 5 KHz First, Then Sham and Then TENS
Started | 8 | 8 | 8 | 7 | 7
Completed | 8 | 8 | 8 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | 5 KHz First, Then TENS and Then Sham | TENS First, Then 5 KHz and Then Sham | Sham First, Then TENS and Then 5KHz | TENS First, Then Sham and Then 5KHz | 5 KHz First, Then Sham and Then TENS
Started | 8 | 8 | 8 | 7 | 7
Completed | 8 | 8 | 8 | 7 | 7
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants who were randomized to receive either 5 KHz, TENS or Sham Stimulation
Arm/Group | All Participants
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.4 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Mechanical Pain Threshold During Treatment
Description: The pressure pain threshold will be measured by a pressure algometer and will be expressed in Newton
Time Frame: during treatment at 15 min
Measure: Mean (Standard Deviation); unit: N
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
N | 57.5 (2.2) | 63.2 (3.1) | 53.8 (2.0)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p < 0.001, ANOVA — A priori threshold for statistical significance. p<0.05

2. Primary Outcome: Thermal Pain Threshold During Treatment
Description: The heat pain threshold will be measured by a computer controlled thermo-foil heating device and will be expressed in ºC
Time Frame: during treatment at 15 min.
Measure: Mean (Standard Deviation); unit: ºC
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
ºC | 57.48 (2.15) | 63.16 (3.08) | 53.82 (2.00)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p = 0.04, ANOVA — A priori threshold for statistical significance. p<0.05

3. Primary Outcome: Nerve Conduction Latency Immediately After Treatment
Description: The compound action potential latencies will be measured and will be expressed in ms.
Time Frame: immediately after treatment at 20 min.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
ms | 3.71 (0.04) | 3.68 (0.04) | 3.63 (0.04)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p = 0.9, ANOVA — A priori threshold for statistical significance. p<0.05

4. Primary Outcome: Tactile Threshold During Treatment
Description: The tactile threshold will be measured with Von Frey filaments and will be expressed in millinewton
Time Frame: during treatment at 15 min.
Measure: Mean (Standard Deviation); unit: mN
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
mN | 18.3 (4.9) | 74.5 (10.3) | 1.1 (0.9)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p = 0.001, ANOVA — A priori threshold for statistical significance. p<0.05

5. Secondary Outcome: Habituation to Electrical Stimulation
Description: The habituation to electrical stimulation along experimental session will be measured by recording the difference on current intensity (mA) at the start of the treatment session (1 min) and end of the same (20 min)
Time Frame: Start treatment session (1 min), end treatment session (20 min)
Population: "Sham stimulation" arm was not included in the analysis because for the habituation to the current the increased intensity was measured throughout the session and in the "Sham group" no current was applied
Measure: Mean (Standard Deviation); unit: mA
Arm/Group | 5 KHz | TENS
Number analyzed (Participants) | 38 | 38
mA | 7.7 (3.1) | 5.5 (2.3)
Statistical Analysis 1: Comparison: 5 KHz vs TENS; Test type: Other; p = 0.003, t-test, 2 sided — A priori threshold for statistical significance. p<0.05

6. Secondary Outcome: Perception Current Comfortability
Description: Participants will choose the current treatment that has found more comfortable
Time Frame: At the end of the third experimental session, 3 days
Population: "Sham stimulation" arm was not included in the analysis of perception current comfortability because in the Sham group no current was applied.
Measure: Count of Participants; unit: Participants
Arm/Group | 5 KHz | TENS
Number analyzed (Participants) | 38 | 38
Participants | 26 | 12
Statistical Analysis 1: Comparison: 5 KHz vs TENS; Test type: Other; p = 0.023, Chi-squared — A priori threshold for statistical significance. p<0.05

7. Secondary Outcome: Change Current Density (mA/cm2)
Description: Change in current density (mA/cm2), it will be recorded at 1 min. start of the treatment session and at 20 min of the same.
Time Frame: at 1 min. treatment session, at 20 min. treatment session
Population: "Sham stimulation" arm was not included in the analysis of "change current density" because in the Sham group no current was applied.
Measure: Mean (Standard Deviation); unit: mA/cm2
Arm/Group | 5 KHz | TENS
Number analyzed (Participants) | 38 | 38
mA/cm2 | 0.62 (0.25) | 0.44 (0.19)
Statistical Analysis 1: Comparison: 5 KHz vs TENS; Test type: Other; p = 0.003, t-test, 2 sided — A priori threshold for statistical significance. p<0,05

8. Secondary Outcome: Change From Baseline in Nerve Conduction Amplitude ( µV)
Description: The compound action potential amplitudes ( µV) will be measured.
Time Frame: Baseline,immediately after treatment at 20 min..
Measure: Mean (Standard Error); unit: µV
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
µV | -0.09 (0.01) | 0.03 (0.02) | -0.4 (0.15)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p = 0.8, ANOVA — A priori threshold for statistical significance. p<0.05

9. Secondary Outcome: Baseline Mechanical Pain Threshold
Description: The pressure pain threshold will be measured by a pressure algometer and will be expressed in Newton
Time Frame: Baseline at 0 min.
Measure: Mean (Standard Deviation); unit: N
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
N | 48.4 (1.7) | 48.3 (1.7) | 54.0 (1.9)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p = 0.02, ANOVA — A priori threshold for statistical significance. p<0.05

10. Secondary Outcome: Mechanical Pain Threshold Post-treatment 20 Min.
Description: The pressure pain threshold will be measured by a pressure algometer and will be expressed in Newton
Time Frame: at 20 min. post-treatment
Measure: Mean (Standard Deviation); unit: N
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
N | 53.8 (1.8) | 55.2 (1.7) | 51.5 (1.8)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p = 0.4, ANOVA — A priori threshold for statistical significance. p<0.05

11. Secondary Outcome: Mechanical Pain Threshold Post-treatment 40 Min.
Description: The pressure pain threshold will be measured by a pressure algometer and will be expressed in Newton.
Time Frame: at 40 min. post-treatment
Measure: Mean (Standard Deviation); unit: N
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
N | 52.0 (2.1) | 52.6 (1.8) | 51.0 (1.7)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p = 0.8, ANOVA

12. Secondary Outcome: Baseline Thermal Pain Threshold
Description: as for outcome 2
Time Frame: Baseline at 0 min.
Measure: Mean (Standard Deviation); unit: ºC
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
ºC | 44.9 (0.4) | 45.0 (0.3) | 44.8 (0.3)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p = 1.0, ANOVA — A priori threshold for statistical significance. p<0.05

13. Secondary Outcome: Thermal Pain Threshold Post-treatment 20 Min.
Description: as for outcome 2
Time Frame: at 20 min. post-treatment
Measure: Mean (Standard Deviation); unit: ºC
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
ºC | 45.1 (0.4) | 45.4 (0.4) | 45.0 (0.4)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p = 0.4, ANOVA — A priori threshold for statistical significance. p<0.05

14. Secondary Outcome: Thermal Pain Threshold Post-treatment 40 Min.
Description: as for outcome 2
Time Frame: at 40 min. post-treatment
Measure: Mean (Standard Deviation); unit: ºC
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
ºC | 45.2 (0.3) | 45.7 (0.3) | 45.2 (0.4)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p = 0.1, ANOVA — A priori threshold for statistical significance. p<0.05

15. Secondary Outcome: Baseline Nerve Conduction Latency
Description: The compound action potential latencies will be measured and will be expressed in ms.
Time Frame: Baseline at 0 min.
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
ms | 3.6 (0.04) | 3.6 (0.04) | 3.6 (0.03)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p = 0.9, ANOVA — A priori threshold for statistical significance. p<0.05

16. Secondary Outcome: Nerve Conduction Latency Post-treatment 20 Min.
Description: The compound action potential latencies will be measured and will be expressed in ms.
Time Frame: at 20 min. post-treatment
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
ms | 3.7 (0.5) | 3.7 (0.5) | 3.7 (0.4)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p = 0.9, ANOVA — A priori threshold for statistical significance. p<0.05

17. Secondary Outcome: Nerve Conduction Latency Post-treatment 40 Min.
Description: The compound action potential latencies will be measured and will be expressed in ms.
Time Frame: at 40 min. post-treatment
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
ms | 3.7 (0.5) | 3.7 (0.4) | 3.6 (0.4)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p = 0.5, ANOVA — A priori threshold for statistical significance. p<0.05

18. Secondary Outcome: Baseline Tactile Threshold
Description: The tactile threshold will be measured with Von Frey filaments and will be expressed in millinewton
Time Frame: Baseline at 0 min.
Measure: Mean (Standard Deviation); unit: mN
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
mN | 1.1 (0.08) | 1.0 (0.00) | 1.0 (0.00)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p = 0.6, ANOVA — A priori threshold for statistical significance. p<0.05

19. Secondary Outcome: Tactile Threshold Post-treatment 20 Min.
Description: The tactile threshold will be measured with Von Frey filaments and will be expressed in millinewton
Time Frame: at 20 min. post-treatment
Measure: Mean (Standard Deviation); unit: mN
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
mN | 1.4 (0.16) | 1.5 (0.2) | 1.0 (0.02)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p = 0.1, ANOVA — A priori threshold for statistical significance. p<0.05

20. Secondary Outcome: Tactile Threshold Post-treatment 40 Min.
Description: The tactile threshold will be measured with Von Frey filaments and will be expressed in millinewton
Time Frame: at 40 min. post-treatment
Measure: Mean (Standard Deviation); unit: mN
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
mN | 1.3 (0.1) | 1.1 (0.08) | 1.0 (0.02)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p = 0.2, ANOVA — A priori threshold for statistical significance. p<0.05

21. Other Pre Specified Outcome: Skin Temperature
Description: Skin temperature (ºC) will be recorded in all assessment times.
Time Frame: Baseline, during treatment at 15 min., immediately after treatment at 20 min., at 20 min. post-treatment, at 40 min. post-treatment
Measure: Mean (Standard Deviation); unit: ºC
Arm/Group | 5 KHz | TENS | Sham Stimulation
Number analyzed (Participants) | 38 | 38 | 38
ºC | 31.3 (0.18) | 31.4 (0.19) | 31.3 (0.2)
Statistical Analysis 1: Comparison: 5 KHz vs TENS vs Sham Stimulation; Test type: Other; p = 1.0, ANOVA — A priori threshold for statistical significance. p<0.05

ADVERSE EVENTS:
Arm/Group | 5 KHz | TENS | Sham Stimulation
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 0/38 | 0/38 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes